CLINICAL TRIAL: NCT01520597
Title: Multicentric Observational NAtional Study on LISteriosis and ListeriA
Brief Title: National Study on Listeriosis and Listeria
Acronym: MONALISA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Pasteur (Industry); French National sanitory (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 09068
Record Dates: First submitted 2012-01-03; First posted 2012-01-30 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Listeriosis; Pregnancy Complications; Infectious; Central Nervous System Infections; Septicemia; Sepsis; Listeria Monocytogenes
Keywords: Multicentric; National; Prospective on; Listeriosis; Listeria
MeSH Terms: conditions — Listeriosis; Pregnancy Complications; Communicable Diseases; Central Nervous System Infections; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Patient with culture-proven listeriosis
- Control: Patient above the age of 18 years with medical background and clinical features compatible with one of the 3 forms of systemic listeriosis: febrile pregnant women (temp > 38°C), febrile patient with co-morbidity for septicaemic listeriosis, and any febrile symptom leading to empiric amoxicillin prescription.

SUMMARY:
Listeriosis is a foodborne infection responsible for severe disease. Three main forms are described: septicaemia, central nervous system infections and maternal-fetal infections. Available data on the disease, are mostly retrospective and do not provide an accurate picture of the clinical / biological / genetic risk factors for the disease, nor identify any element to determine which patients are at higher risk of death, severe neurological impairment or fetal loss.

The primary purpose of the study is to identify clinical, biological and genetic risk factors for systemic listeriosis and the determinants of listeriosis-associated mortality in the setting of a large prospective nation-wide study.

DETAILED DESCRIPTION:
Context: Listeriosis is a foodborne infection responsible for severe disease. Surveillance of human listeriosis in France is based on both mandatory reporting of cases and voluntary submission of L. monocytogenes strains to the National Reference Center for Listeria (NRC) since 1999. The exhaustiveness of this reporting estimated by capture-recapture is of at least 87%. A recent and consistent increase of sporadic and cluster-associated systemic listeriosis cases has been reported in Europe since several years (since 2006 in France), but remains poorly understood in the absence of any new environmental risk factor(s). A total of 322 cases have been reported in 2009 in France. Three main clinical forms are identified: septicemia, central nervous system and maternal-fetal infection. They have been characterized only through retrospective studies and pooling of heterogeneous patients. Such studies do not provide an accurate picture of the disease and fail to identify precise biological / genetic risk factors for the disease. Prognostic factors associated with higher risk of death, of severe neurological impairment or of fetal loss also remain to be determined.

Main purpose:

- to study clinical, biological and genetic risk factors for systemic listeriosis and identify determinants of listeriosis-associated mortality in the setting of a large prospective nation-wide study

Secondary purposes:

* to determine the clinical/biological and radiological presentation of listeriosis
* to describe and further study current therapeutic practices in the 3 forms of the disease (namely, septicaemic, neurologic and maternal-fetal)
* to identify inherited risk factors for listeriosis

Ancillary studies:

- to evaluate serologic/PCR diagnostic tools

Study design:

National prospective multicenter study with nested case control study. Clinical, biological and radiological data are collected. Additionally a questionnaire focusing on dietary habits is proposed. A bank of biological samples is performed. For each patient, 25ml of heparinized blood / and 2ml of serum are collected per patient

ELIGIBILITY:
Inclusion Criteria:

Case:

* Patient with culture-proven listeriosis (blood, CSF, fetal/placental sample, other…).

Control:

* Patient above the age of 18 years with medical background and clinical features compatible with one of the 3 forms of systemic listeriosis: febrile pregnant women (temp > 38°C), febrile patient with co-morbidity for septicaemic listeriosis, and any febrile symptom leading to empiric amoxicillin prescription.
* For feasibility reasons, controls are included in Paris (France) emergency wards.

Exclusion Criteria:

Case:

* Patient who would refuse to sign informed consent agreement

Control:

* Patient who would refuse to sign informed consent agreement, or whose samples would evidence L. monocytogenes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Case: patient with culture-proven listeriosis (blood CSF, fetal/placental sample, other…).
  Controls: patient above the age of 18 years with medical background and clinical features compatible with one of the 3 forms of systemic listeriosis: febrile pregnant women (temp > 38°C), febrile patient with co-morbidity for septicaemic listeriosis, and any febrile symptom leading to empiric amoxicillin prescription.
Sampling Method: Non-Probability Sample
Enrollment: 2132 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2013-04-05 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Clinical, biological and genetic risk factors for systemic listeriosis | At Day 1 (case and control)
  Clinical, biological and genetic risk factors for systemic listeriosis and identify determinants of listeriosis-associated mortality in the setting of a large prospective nation-wide study
Clinical, biological and genetic risk factors for systemic listeriosis | At Day 90 (case)
  Clinical, biological and genetic risk factors for systemic listeriosis and identify determinants of listeriosis-associated mortality in the setting of a large prospective nation-wide study

SECONDARY OUTCOMES:
Clinical/biological and radiological presentation of listeriosis | At Day 1 and Day 90 (case), at Day 1 (control)
  To determine the clinical/biological and radiological presentation of listeriosis
Current therapeutic practices | At Day 1 and Day 90 (case), at Day 1 (control)
  to describe and further study current therapeutic practices in the 3 forms of the disease (septicaemic, neurological and maternal-fetal)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Charlier, MD, PhD, Principal Investigator — Institut Pasteur; Lecuit Marc, MD, PhD, Study Director — Institut Pasteur
Locations (1):
- Centre National de Reference et Centre Collaborateur OMS Listeria, Institut Pasteur, Paris, France

REFERENCES:
- [Background] Mylonakis E, Hohmann EL, Calderwood SB. Central nervous system infection with Listeria monocytogenes. 33 years' experience at a general hospital and review of 776 episodes from the literature. Medicine (Baltimore). 1998 Sep;77(5):313-36. doi: 10.1097/00005792-199809000-00002. PMID 9772921
- [Background] Mylonakis E, Paliou M, Hohmann EL, Calderwood SB, Wing EJ. Listeriosis during pregnancy: a case series and review of 222 cases. Medicine (Baltimore). 2002 Jul;81(4):260-9. doi: 10.1097/00005792-200207000-00002. No abstract available. PMID 12169881
- [Background] Lecuit M, Vandormael-Pournin S, Lefort J, Huerre M, Gounon P, Dupuy C, Babinet C, Cossart P. A transgenic model for listeriosis: role of internalin in crossing the intestinal barrier. Science. 2001 Jun 1;292(5522):1722-5. doi: 10.1126/science.1059852. PMID 11387478
- [Background] Disson O, Grayo S, Huillet E, Nikitas G, Langa-Vives F, Dussurget O, Ragon M, Le Monnier A, Babinet C, Cossart P, Lecuit M. Conjugated action of two species-specific invasion proteins for fetoplacental listeriosis. Nature. 2008 Oct 23;455(7216):1114-8. doi: 10.1038/nature07303. Epub 2008 Sep 17. PMID 18806773
- [Background] Charlier C, Leclercq A, Cazenave B, Desplaces N, Travier L, Cantinelli T, Lortholary O, Goulet V, Le Monnier A, Lecuit M; L monocytogenes Joint and Bone Infections Study Group. Listeria monocytogenes-associated joint and bone infections: a study of 43 consecutive cases. Clin Infect Dis. 2012 Jan 15;54(2):240-8. doi: 10.1093/cid/cir803. Epub 2011 Nov 18. PMID 22100574
- [Result] Charlier C, Perrodeau E, Leclercq A, Cazenave B, Pilmis B, Henry B, Lopes A, Maury MM, Moura A, Goffinet F, Dieye HB, Thouvenot P, Ungeheuer MN, Tourdjman M, Goulet V, de Valk H, Lortholary O, Ravaud P, Lecuit M; MONALISA study group. Clinical features and prognostic factors of listeriosis: the MONALISA national prospective cohort study. Lancet Infect Dis. 2017 May;17(5):510-519. doi: 10.1016/S1473-3099(16)30521-7. Epub 2017 Jan 28. PMID 28139432
- [Result] Charlier C, Barrault Z, Rousseau J, Kermorvant-Duchemin E, Meyzer C, Semeraro M, Fall M, Coulpier G, Leclercq A, Charles MA, Ancel PY, Lecuit M. Long-term neurological and neurodevelopmental outcome of neonatal listeriosis in France: a prospective, matched, observational cohort study. Lancet Child Adolesc Health. 2023 Dec;7(12):875-885. doi: 10.1016/S2352-4642(23)00195-5. Epub 2023 Oct 20. PMID 37871603
- [Result] Charlier C, Poiree S, Delavaud C, Khoury G, Richaud C, Leclercq A, Helenon O, Lecuit M; MONALISA Study Group. Imaging of Human Neurolisteriosis: A Prospective Study of 71 Cases. Clin Infect Dis. 2018 Oct 15;67(9):1419-1426. doi: 10.1093/cid/ciy449. PMID 29796652
- [Result] Charlier C, Kermorvant-Duchemin E, Perrodeau E, Moura A, Maury MM, Bracq-Dieye H, Thouvenot P, Vales G, Leclercq A, Ravaud P, Lecuit M. Neonatal Listeriosis Presentation and Outcome: A Prospective Study of 189 Cases. Clin Infect Dis. 2022 Jan 7;74(1):8-16. doi: 10.1093/cid/ciab337. PMID 33876229
- [Result] Charlier C, Perrodeau E, Levallois C, Cachina T, Dommergues M, Salomon LJ, Azria E, Goffinet F, Ravaud P, Lecuit M. Causes of fever in pregnant women with acute undifferentiated fever: a prospective multicentric study. Eur J Clin Microbiol Infect Dis. 2020 May;39(5):999-1002. doi: 10.1007/s10096-019-03809-3. Epub 2020 Jan 18. PMID 31955353